CLINICAL TRIAL: NCT05139511
Title: Analysis of the Efficacy and Safety of Intense Pulsed Light Treatment for the Ocular Surface in Patients Who Will Undergo Laser Refractive Surgery
Brief Title: Analysis of the Results of Intense Pulsed Light Treatment Previously to Laser Refractive Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vissum, Instituto Oftalmológico de Alicante (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPL-2020
Record Dates: First submitted 2021-11-04; First posted 2021-12-01 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Meibomian Gland Dysfunction; Blepharitis
Keywords: Intense pulsed light; LASIK / SMILE
MeSH Terms: conditions — Meibomian Gland Dysfunction; Blepharitis; Smiling | interventions — Intense Pulsed Light Therapy; Control Groups

STUDY DESIGN:
Intervention Model Description: Clinical experimental controlled trial, double-blind in which participants will be randomized into 2 groups: a study group and a control group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): IPL + laser refractive surgery
  Interventions: Device: Study group
- Control group (Placebo Comparator): Laser refractive surgery without IPL
  Interventions: Other: Control group

INTERVENTIONS:
Device: Study group — The IPL therapy consists in a polychromatic pulses of light not coherent and not collimated. The therapy leads to a series of processes such as the destruction of superficial blood vessels and thus the reduction of local inflammation, the liquefy of the meibum and an antimicrobial, anti-inflammatory and antioxidant effects. The therapy is performed over the cheeks, nose and upper eyelids.
  Other Names: Intense pulsed light therapy (Lumenis M22)
  Arms: Study group
Other: Control group — Same procedure but without energy
  Arms: Control group

SUMMARY:
Dry eye is often reported as the most common complication after a laser refractive surgery. Any refractive procedure can lead an impact on the corneal surface and the tear film.

The main cause of this dry eye is the corneal denervation caused by the destruction of the anterior stromal nerves during the ablative procedure. This loss of corneal sensitivity leads to a decrease in the blink reflex, a decrease in the secretion rate of the meibomian glands and finally an evaporated dry eye. There is also a chronic inflammation at the corneal surface that produces an increase of inflammatory cytokines and a dysfunction of the meibomian glands.

Yu et al have described incidences of dry eye closed to 60% after the first month of LASIK. Hovanesian et al have observed dry eye symptoms in 50% of patients 6 months after surgery. Donnenfeld et al describe 15% of moderate dry eye in the following 3 months and 5% of severe dry eye in the first 6 months. A small number of patients will present with chronic dry eye symptoms for more than 1 year. Bower et al analyzed its incidence in 0.8% Alterations in the tear film also decrease the quality of the retinal image and produce greater number of high-order due to the irregular.

Pulsed light therapy (IPL) applied preoperatively in patients who undergo a laser refractive surgery may prevent the post-surgical dry eye and improve the refractive results. The aim of our study is to evaluate the usefulness of the applied therapy for the prevention of dry eye in patients that undergo a corneal refractive procedure.

DETAILED DESCRIPTION:
1. Design Clinical experimental controlled trial, double-blind in which participants will be randomized into 2 groups: a study group (IPL + laser refractive surgery) and a control group (laser refractive surgery without IPL).

   The study will be conducted in accordance with Law 14/2007 of 3 July, on Biomedical Research, the Declaration of Helsinki (October 2013 version), standards of Good Clinical Practice and legislation in this area.

   All participants included in the study should read the Information Sheet and sign the informed and voluntary consent.
2. Participants Participants from Vissum Clinic that present the inclusion criteria and none of the exclusion criteria.

   The investigators will start the study with a preliminary project and depending on the results obtained, the investigators will apply these values to calculate the final sample size using the T-student-Fischer test for unilateral hypotheses and for a type 1 or α error of 5%. and a type 2 or β error of 20%.
3. Parameters evaluated Primary measures: age, sex, skin phototype, visual acuity with and without correction, refraction, cycloplegic refraction, OSDI and VAS questionnaire, use of artificial tears, oxford scale, lacrimal meniscus height, tear break-up time, conjunctival hyperemia, meibography and slit lamp examination.

   Secondary measures: corneal topography and tomography (MS-39, CSO, Italy), corneal aberrometry (MS-39, CSO, Italy), ocular aberrometry (Osiris, CSO, Italy), analysis of contrast sensitivity (CSV-1000, Vector vision), photographic capture of the epithelial defect in PRK, pre-surgical and postsurgical photographic capture of the eyelid changes in PRK.

   The measurement of the different objective variables will be carried out in the clinic. The measurement of the subjective variables will be carried out by two ophthalmologists, both masked.
4. Surgery and follow-up Participants who are candidates for a LASIK or SMILE procedure will receive, after randomization, IPL treatment in both eyes (experimental group) or sham IPL (control group). In the case of participant candidate for a PRK procedure, an intra-subject control group will be used, where one eye will receive the IPL treatment (right eyes) and the left contralateral eye the sham IPL treatment (control).

   Refractive surgeries will be performed exclusively two ophthalmologists following the same surgical protocol.

   IPL therapy (M22, Lumenis LTD, Israel) will be performed following the same protocol (standardized facial and periocular application with automatically adjusted energy according to Fitzpatrick skin classification). Three IPL sessions will be applied (simulated in the case of the control group): 7 days before the intervention, 7 days after the intervention, and 30 days after the intervention. The total postsurgical follow-up will be 6 months.
5. Statistical analyses All demographic and clinical data will be collected in a database and analyzed with the SPSS statistical package for Windows version 22.0. A p <0.05% will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age who are undergoing a corneal laser refractive surgery after a medical indication by the Vissum ophthalmologist

Exclusion Criteria:

* Pregnancy
* Piercings
* Fitzpatrick skin classification V and VI
* Autoimmune diseases
* Epilepsy
* Previous history of herpes or ocular pathology
* Pathological or suspicious corneal topography
* Treatment in the previous month with corticosteroids, antihistamines or topical vasoconstrictors.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
OSDI questionnaire | 0 day
  It measures the severity of ocular surface symptoms and includes 12 items organized into 3 subscales; eye discomfort, functionality and environmental factors. After completing the questionnaire, a final score is obtained that when it is higher than 13 indicates ocular surface pathology.
Change from Baseline OSDI questionnaire | 7 day
  It measures the severity of ocular surface symptoms and includes 12 items organized into 3 subscales; eye discomfort, functionality and environmental factors. After completing the questionnaire, a final score is obtained that when it is higher than 13 indicates ocular surface pathology.
Change from Baseline OSDI questionnaire | 30 day
  It measures the severity of ocular surface symptoms and includes 12 items organized into 3 subscales; eye discomfort, functionality and environmental factors. After completing the questionnaire, a final score is obtained that when it is higher than 13 indicates ocular surface pathology.
Change from Baseline OSDI questionnaire | 90 day
  It measures the severity of ocular surface symptoms and includes 12 items organized into 3 subscales; eye discomfort, functionality and environmental factors. After completing the questionnaire, a final score is obtained that when it is higher than 13 indicates ocular surface pathology.
Change from Baseline OSDI questionnaire | 180 day
  It measures the severity of ocular surface symptoms and includes 12 items organized into 3 subscales; eye discomfort, functionality and environmental factors. After completing the questionnaire, a final score is obtained that when it is higher than 13 indicates ocular surface pathology.
Lacrimal meniscus height | 0 day
  Measured in millimeters by Ocular Keratograph 5M, a value greater than 0.20 mm is considered normal
Change from Baseline Lacrimal meniscus height | 7 day
  Measured in millimeters, a value greater than 0.20 mm is considered normal
Change from Baseline Lacrimal meniscus height | 30 day
  Measured in millimeters, a value greater than 0.20 mm is considered normal
Change from Baseline Lacrimal meniscus height | 90 day
  Measured in millimeters, a value greater than 0.20 mm is considered normal
Change from Baseline Lacrimal meniscus height | 180 day
  Measured in millimeters, a value greater than 0.20 mm is considered normal
Tear Break-up-time | 0 day
  Time elapsed from the last blink to the appearance of the first tear discontinuity measured by Ocular Keratograph 5M. A title longer than 5 seconds is considered normal.
Change from Baseline Tear Break-up-time | 7 day
  time elapsed from the last blink to the appearance of the first tear discontinuity measured by Ocular Keratograph 5M. A title longer than 5 seconds is considered normal.
Change from Baseline Tear Break-up-time | 30 day
  time elapsed from the last blink to the appearance of the first tear discontinuity measured by Ocular Keratograph 5M. A title longer than 5 seconds is considered normal.
Change from Baseline Tear Break-up-time | 90 day
  time elapsed from the last blink to the appearance of the first tear discontinuity measured by Ocular Keratograph 5M. A title longer than 5 seconds is considered normal.
Change from Baseline Tear Break-up-time | 180 day
  time elapsed from the last blink to the appearance of the first tear discontinuity measured by Ocular Keratograph 5M. A title longer than 5 seconds is considered normal.
Conjunctival and ciliary hyperemia. | 0 day
  Grade of red eye measured by Ocular Keratograph 5M. Jenvis ranking from 0 to 4 (normal, mild, moderate, severe)
Change from Baseline Conjunctival and ciliary hyperemia. | 7 day
  Grade of red eye measured by Ocular Keratograph 5M. Jenvis ranking from 0 to 4 (normal, mild, moderate, severe)
Change from Baseline Conjunctival and ciliary hyperemia. | 30 day
  Grade of red eye measured by Ocular Keratograph 5M. Jenvis ranking from 0 to 4 (normal, mild, moderate, severe)
Change from Baseline Conjunctival and ciliary hyperemia. | 90 day
  Grade of red eye measured by Ocular Keratograph 5M. Jenvis ranking from 0 to 4 (normal, mild, moderate, severe)
Change from Baseline Conjunctival and ciliary hyperemia. | 180 day
  Grade of red eye measured by Ocular Keratograph 5M. Jenvis ranking from 0 to 4 (normal, mild, moderate, severe)
Upper and lower meibography | 0 day
  Measured by Oculus Keratograph 5M. Observes and evaluates morphological changes of the meibomian glands Meiboscore classification
  * Grade 0: no loss of meibomian glands.
  * Grade 1: loss of less than 1/3 of the total surface of the meibomian glands.
  * Grade 2: loss of 1/3 to 2/3 of the total area.
  * Grade 3: loss of more than 2/3 of the surface.
Change from Baseline Upper and lower meibography | 7 day
  Measured by Oculus Keratograph 5M. Observes and evaluates morphological changes of the meibomian glands Meiboscore classification
  * Grade 0: no loss of meibomian glands.
  * Grade 1: loss of less than 1/3 of the total surface of the meibomian glands.
  * Grade 2: loss of 1/3 to 2/3 of the total area.
  * Grade 3: loss of more than 2/3 of the surface.
Change from Baseline Upper and lower meibography | 30 day
  Measured by Oculus Keratograph 5M. Observes and evaluates morphological changes of the meibomian glands Meiboscore classification
  * Grade 0: no loss of meibomian glands.
  * Grade 1: loss of less than 1/3 of the total surface of the meibomian glands.
  * Grade 2: loss of 1/3 to 2/3 of the total area.
  * Grade 3: loss of more than 2/3 of the surface.
Change from Baseline Upper and lower meibography | 90 day
  Measured by Oculus Keratograph 5M. Observes and evaluates morphological changes of the meibomian glands Meiboscore classification
  * Grade 0: no loss of meibomian glands.
  * Grade 1: loss of less than 1/3 of the total surface of the meibomian glands.
  * Grade 2: loss of 1/3 to 2/3 of the total area.
  * Grade 3: loss of more than 2/3 of the surface.
Change from Baseline Upper and lower meibography | 180 day
  Measured by Oculus Keratograph 5M. Observes and evaluates morphological changes of the meibomian glands Meiboscore classification
  * Grade 0: no loss of meibomian glands.
  * Grade 1: loss of less than 1/3 of the total surface of the meibomian glands.
  * Grade 2: loss of 1/3 to 2/3 of the total area.
  * Grade 3: loss of more than 2/3 of the surface.

SECONDARY OUTCOMES:
Visual acuity | 0 day
  Visual acuity with and without correction, measured on a decimal scale, determined by the Snellen panel, placing the examined person at a distance of 6 meters, will be collected by an optician.
Change from Baseline Visual acuity | 180 day
  Visual acuity with and without correction, measured on a decimal scale, determined by the Snellen panel, placing the examined person at a distance of 6 meters, will be collected by an optician.
Corneal topography | 0 day
  Performs an analysis of the cornea, which allows evaluating the shape and quantifying the power of the different curvatures
Change from Baseline Corneal topography | 180 day
  Performs an analysis of the cornea, which allows evaluating the shape and quantifying the power of the different curvatures
Corneal aberrometry | 0 day
  Technique that analyzes complex systems of light waves to quantify the set of optical aberrations that exist within the ocular structure.
Change from Baseline Corneal aberrometry | 180 day
  Technique that analyzes complex systems of light waves to quantify the set of optical aberrations that exist within the ocular structure.
Analysis of contrast sensitivity | 0 day
  Contrast Sensitivity is a test that assesses a person's ability to identify an object and separate it from the background Contrast sensitivity is evaluated with charts that can be used as projected or wall acuity charts.
Change from Baseline Analysis of contrast sensitivity | 180 day
  Contrast Sensitivity is a test that assesses a person's ability to identify an object and separate it from the background Contrast sensitivity is evaluated with charts that can be used as projected or wall acuity charts.
VAS questionnaire | 0 day
  investigates the intensity of the ocular surface symptoms from 0 to 100 (normal- severe)
Change from Baseline VAS questionnaire | 180 day
  investigates the intensity of the ocular surface symptoms from 0 to 100 (normal- severe)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Alió del Barrio, MD, PhD, Principal Investigator — Vissum Miranza; Maria Martinez Hergueta, MD, Study Chair — Universidad Miguel Hernández; Maria A Amesty, MD, PhD, Study Chair — Vissum Miranza; Mario Cantó Cerdan, MSc, Study Chair — Vissum Miranza; Alejandra Rodriguez, MSc, PhD, Study Chair — Vissum Miranza; Jorge L Alió y Sanz, MD, PhD, Study Chair — Vissum Miranza
Locations (1):
- Alicante Vissum Miranza, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be anonymized by assigning a code file and only authorized personnel will have access to personally identifiable data. The highest levels of professional conduct and confidentiality will always be maintained, complying with Organic Law 3/2018, of December 5, on the Protection of Personal Data and guarantee of digital rights.

REFERENCES:
- [Result] Solomon R, Donnenfeld ED, Perry HD. The effects of LASIK on the ocular surface. Ocul Surf. 2004 Jan;2(1):34-44. doi: 10.1016/s1542-0124(12)70022-8. PMID 17216074
- [Result] Toda I. Dry Eye After LASIK. Invest Ophthalmol Vis Sci. 2018 Nov 1;59(14):DES109-DES115. doi: 10.1167/iovs.17-23538. PMID 30481814
- [Result] Ge J, Liu N, Wang X, Du Y, Wang C, Li Z, Li J, Wang L. Evaluation of the efficacy of optimal pulsed technology treatment in patients with cataract and Meibomian gland dysfunction in the perioperative period. BMC Ophthalmol. 2020 Mar 18;20(1):111. doi: 10.1186/s12886-020-01357-5. PMID 32188437
- [Result] Jung JW, Han SJ, Nam SM, Kim TI, Kim EK, Seo KY. Meibomian gland dysfunction and tear cytokines after cataract surgery according to preoperative meibomian gland status. Clin Exp Ophthalmol. 2016 Sep;44(7):555-562. doi: 10.1111/ceo.12744. Epub 2016 May 1. PMID 26989003
- [Result] Yu EY, Leung A, Rao S, Lam DS. Effect of laser in situ keratomileusis on tear stability. Ophthalmology. 2000 Dec;107(12):2131-5. doi: 10.1016/s0161-6420(00)00388-2. PMID 11097583
- [Result] Hovanesian JA, Shah SS, Maloney RK. Symptoms of dry eye and recurrent erosion syndrome after refractive surgery. J Cataract Refract Surg. 2001 Apr;27(4):577-84. doi: 10.1016/s0886-3350(00)00835-x. PMID 11311627
- [Result] Nettune GR, Pflugfelder SC. Post-LASIK tear dysfunction and dysesthesia. Ocul Surf. 2010 Jul;8(3):135-45. doi: 10.1016/s1542-0124(12)70224-0. PMID 20712970
- [Result] Cote S, Zhang AC, Ahmadzai V, Maleken A, Li C, Oppedisano J, Nair K, Busija L, Downie LE. Intense pulsed light (IPL) therapy for the treatment of meibomian gland dysfunction. Cochrane Database Syst Rev. 2020 Mar 18;3(3):CD013559. doi: 10.1002/14651858.CD013559. PMID 32182637
- [Result] Rong B, Tang Y, Tu P, Liu R, Qiao J, Song W, Toyos R, Yan X. Intense Pulsed Light Applied Directly on Eyelids Combined with Meibomian Gland Expression to Treat Meibomian Gland Dysfunction. Photomed Laser Surg. 2018 Jun;36(6):326-332. doi: 10.1089/pho.2017.4402. Epub 2018 Apr 24. PMID 29688838